CLINICAL TRIAL: NCT05330065
Title: A Phase Ib/II Study of Intrapleural Administration of Bevacizumab and Camrelizumab for Patients With Malignant Pleural Effusion
Brief Title: A Study of Intrapleural Administration of Bevacizumab and Camrelizumab for Malignant Pleural Effusion
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: The First Affiliated Hospital of Zhengzhou University (Other)
Responsible Party: Principal Investigator, Feng Wang, Chief Physician, The First Affiliated Hospital of Zhengzhou University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SHR-1210-MPE-001
Record Dates: First submitted 2022-02-06; First posted 2022-04-15 (Actual); Last update posted 2022-04-15 (Actual); Status verified 2022-04

CONDITIONS: Malignant Pleural Effusion
MeSH Terms: conditions — Pleural Effusion, Malignant | interventions — Bevacizumab; camrelizumab

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Bevacizumab and Camrelizumab for Malignant Pleural Effusion (Experimental)
  Interventions: Drug: bevacizumab and camrelizumab

INTERVENTIONS:
Drug: bevacizumab and camrelizumab — Stage 1 was classical "3+3" dose escalation with pts assigned to one of the following 3 cohorts, Cohort A:Avastin 5mg/kg once every 2 weeks and camrelizumab 100mg once every 2 weeks;Cohort B:Avastin 7.5mg/kg once every 2 weeks and camrelizumab 100mg once every 2 weeks;Cohort C:Avastin 7.5mg/kg once every 2 weeks and camrelizumab 200mg once every 2 weeks.DLT was observed for 28 days.

SUMMARY:
Patients with a variety of malignancies can develop malignant pleural effusion (MPE). MPE can cause significant symptoms and result in a marked decrease in quality of life and a poor prognosis. MPE is primarily considered as an immune and vascular manifestation of pleural metastases. The combined use of anti-angiogenic therapy and immunotherapy may be a promising strategy for MPE.

This is a Phase Ib/II clinical trial to evaluate the safety and tolerability of administering bevacizumab and camrelizumab into the intrapleural space of subjects with malignant pleural effusion through a pleurX catheter.

DETAILED DESCRIPTION:
This study is a phase Ib/II, single arm study with main purpose to evaluate the safety, tolerability and efficacy of intrapleural administration of bevacizumab and camrelizumab in subjects with malignant pleural effusion.

The study aims to recruit 9 - 15 subjects in phase 1, and once the safety, tolerability and the preliminary efficacy of bevacizumab and camrelizumab reach an optimal target exposure for recommended dose (RD), phase 2a will be opened for enrolment of approximately 40 subjects

ELIGIBILITY:
Inclusion Criteria:

1. Be ≥ 18 years of age on day of signing informed consent.
2. Histologically or cytologically documented malignant pleural effusion
3. Histologically confirmed cancer
4. Malignant pleural effusion clinically judged as not responsive to conventional systemic therapy(ies) for primary malignancy
5. Adequate liver and renal function as defined below:
6. Eastern Cooperative Oncology Group (ECOG) performance status ≤ 2
7. Life expectancy of > 12 weeks
8. Willing and able to provide written, signed informed consent after the nature of the study has been explained, and prior to any research-related procedures
9. Females of childbearing potential must have a negative serum pregnancy test at screening and be willing to have additional serum pregnancy tests during the study.
10. Willing and able to comply with all study procedures

Exclusion Criteria：

1. Receiving any investigational agent, or using an investigational device, currently or within 28 days or 5 half-lives of Day 1 of treatment on this study, whichever is longer.
2. Has had prior chemotherapy, targeted small molecule therapy, or radiation therapy within 2 weeks prior to study Day 1.
3. Has had a prior monoclonal antibody within 4 weeks prior to study Day 1, or who has not recovered to, ≤ Grade 1 toxicity at baselines from adverse events due to agents administered more than 4 weeks earlier.
4. Has received prior intrapleural administration with an anti-programmed cell death receptor (PD)-1, anti-PD-L1, anti-PD-L2, anti-CD137, or anti-Cytotoxic T-lymphocyte-associated antigen-4 (CTLA-4) antibody (including ipilimumab or any other antibody or drug specifically targeting T-cell co-stimulation or checkpoint pathways).
5. Has received prior intrapleural administration with bevacizumab or Endostar.
6. Any concurrent chemotherapy, intraperitoneal (IP), biologic or hormonal therapy for cancer treatment. Concurrent use of hormonal therapy for non-cancer-related conditions (e.g., hormone replacement therapy) is acceptable.
7. Major surgery within 28 days prior to day 1 of study treatment from which the patient has not completely recovered.
8. Has a diagnosis of immunodeficiency or is receiving systemic steroid therapy or any other form of immunosuppressive therapy within 7 days prior to the first dose of trial treatment.
9. Has a history of non-infectious pneumonitis that required steroids; currently active non-infectious pneumonitis; or evidence of interstitial lung disease.
10. Has an active infection requiring systemic therapy or history of uncontrolled infection.
11. Concurrent disease or condition which, in the opinion of the Investigator, would pose a risk to patient safety or interfere with study participation or interpretation of individual patient results
12. Breastfeeding at screening or planning to become pregnant (self or partner) at any time during study participation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Estimated)
Dates: Start 2022-08-01 (Estimated); Primary Completion 2023-08-31 (Estimated); Study Completion 2024-08-31 (Estimated)

PRIMARY OUTCOMES:
Adverse Events (Safety) | up to 12 months
  Incidence of safety events including: adverse events (AEs), Serious AEs, and dose limiting toxicities (DLTs) AEs:Percentage of participants with adverse events; SAEs:Percentage of participants with Serious AEs; Dose limiting toxicity (DLT) is referred to grade 3 non-hematological toxicity or grade 4 hematological toxicity according to NCI CTCAE 4.0 criteria.
ORR | up to 12 months
  Complete remission (CR) was considered when the accumulated fluid had disappeared and was stable for at least four weeks; partial remission (PR) was considered when >50% of the accumulated fluid had disappeared, symptoms had improved, and the remaining fluid had failed to increase for at least four weeks; The total efficiency ORR was calculated by taking the sum of CR+PR

SECONDARY OUTCOMES:
Exploratory biomarkers | up to 12 months
  1. The expression levels of PD-L1 CPS and TPS in baseline Tumor cells embedded in initial pleural fluid sediment
  2. Levels of VEGF and its soluble receptor SVEGFR-1 in pleural fluid and plasma (THE levels of VEGF and SVEGFR-1 in pleural fluid and plasma are determined by ELISA) ;
  3. Flow cytometry is used to detect CD8+ CD69+ cell , CD8+ IFN-G + cell , CD8+ Granzyb + cell and CD8+ PD-1+ in MPE before and after intrathoracic injection of the study drug.;
  4. The release levels of TNF-A and IL-1B in the supernatant of pleural effusion and peripheral blood using ELISA
Quality of life questionnaire EORTC QLQ 30 | up to12 months
  Scale from 1-100 for 30 items, higher score indicates a better situation.

CONTACTS AND LOCATIONS:
Overall Officials: Feng Wang, Principal Investigator — The First Affiliated Hospital of Zhengzhou University